CLINICAL TRIAL: NCT02445430
Title: Genetics of Arteriovenous Malformations
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Translational Genomics Research Institute (Other); The Joe Niekro Foundation (Unknown)
Responsible Party: Principal Investigator, Lisa Arnold, Research Manager, St. Joseph's Hospital and Medical Center, Phoenix
Other Study IDs: 15BN031
Record Dates: First submitted 2015-05-11; First posted 2015-05-15 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Arteriovenous Malformation
MeSH Terms: conditions — Arteriovenous Malformations

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva, blood, tissue (if undergoing AVM resection)
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this study is to identify genetic alterations resulting in the development of arteriovenous malformation (AVM) in the central nervous system.

DETAILED DESCRIPTION:
The study will include AVM patients and members of their nuclear family. All patients will donate a sample of saliva (5 mL) or blood (10 mL). Basic demographic and clinical parameters will be collected, including ethnicity, age at first presentation, symptoms at presentation, history of subsequent symptoms, treatment history, Spetzler-Martin AVM grade, medication history, and other pertinent medical information. In patients undergoing AVM resection, a small sample of the AVM will be collected for concurrent genomic analysis. Family members will donate saliva (5mL) and document their relationship to the patient (i.e., parent, sibling, child, etcl). Nucleic acids will be isolated from the saliva/blood samples, and genetic sequencing will be carried out. When a surgical sample of the AVM is available, nucleic acids will be obtained and transcriptome profiling will be performed. Identification of genetic alterations common to patients with AVM and not present in samples from parents and siblings will greatly aid in identification of pathways associated with AVM formation. Candidate sequences will be chosen by differential expression (p<0.05) and fold-changes. Once identified, mechanisms for the rapid detection of marker sequences will be developed and their predictive value tested in future collections.

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 and 60 years inclusive
* Diagnosis of AVM or nuclear family member of a patient with AVM
* Grants access to saliva, blood, and/or tissue

Exclusion Criteria:

* Age less than 6 years or greater than 61 years
* Nuclear family members who do not share the same parents as the AVM patient

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Male and female persons with AVM and their immediate family members
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Identification of genetic alterations common to patients with AVM | sample analysis will take an expected average of six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zabramski, MD, Principal Investigator — Barrow Neurosurgical Associates
Locations (1):
- Barrow Neurological Institute, Phoenix, Arizona, United States